CLINICAL TRIAL: NCT04816786
Title: Prognostic Factors and Predictors of Mortality in COVID-19 Patients Admitted to the ICU. An Aid for Triage, Counseling, and Resource Allocation
Brief Title: COVID-19 Patients Admitted to the ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Waleed burhamah, Dr. Waleed burhamah, General surgery resident MKH MB BCH BOA, Ministry of Health, Kuwait
Other Study IDs: 1591/2020
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Admitted to ICU and died during the hospital stay.
  Interventions: Other: no intervention will be administered, this is a retrospective observational study.
- Group 2: Admitted to ICU was were discharged.
  Interventions: Other: no intervention will be administered, this is a retrospective observational study.

INTERVENTIONS:
Other: no intervention will be administered, this is a retrospective observational study. — no intervention will be administered, this is a retrospective observational study.

SUMMARY:
A retrospective analysis of the adult COVID-19 patients admitted to the ICU. A chart review will be conducted and multiple baseline characteristics, demographics, and treatments given will be recorded.

Variables collected will include Age, Gender, BMI, Smoking status, Past medical history, Vital signs on admission, symptoms on admission, duration of symptoms, laboratory results on admission, treatment given. Treatment options will include (Steroids, plasma exchange, IVIG, antibiotics, mode of respiratory support).

Primary outcomes will include; Death, duration of ICU stay, duration of mechanical ventilation, in-hospital complications.

A regression model will be used to predict poor prognostic factors. Inclusion criteria: patients with confirmed PCR results for COVID-19 AND require ICU admission. Exclusion criteria: those with negative results, pediatric patients and those not requiring ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Positive PCR test for COVID-19
* Require admission to ICU

Exclusion Criteria:

* Pediatric patients\
* Any patient not requiring admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the hospital and suspected of having the COVID-19 virus. Patients who are positive on a PCR test are usually traiged to be managed on the wards Vs ICU (Intensive care unit). This is based on a number of parameters; including but not limited to The severity of the symptoms, vital signs, lab results, co-morbidities, age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Death | 30 day mortality
  Death Vs No Death
Duration of ICU stay | 30 days
  Duration of ICU stay
Duration of mechanical ventilation | 30 days
  The duration the patient required support from a mechanical ventilator

SECONDARY OUTCOMES:
In-Hospital complications | 30 days
  Wether patients developed in hospital complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Mubarak al Kabeer hospital, Kuwait City, Outside U.S./Canada, Kuwait

IPD SHARING:
Plan to Share IPD: No